CLINICAL TRIAL: NCT06703918
Title: A Retrospective Cohort Study on the Epidemiological Characteristics and Biomarkers of Clostridium Difficile Infection in Infants
Brief Title: Study on Clostridium Difficile Infection in Infants
Status: Recruiting | Type: Observational
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Westlake University (Other)
Responsible Party: Sponsor
Other Study IDs: KY-20240613-0201-01
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; Infants; Epidemiology; Biomarkers
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: This group includes infants and young children diagnosed with Clostridium difficile infection (CDI). Participants in this group have been identified based on medical records andpatient questionnaires showing confirmed CDI diagnosis. This group will be analyzed for epidemiological characteristics and biomarkers associated with CDI.
- Control Group: This group includes infants and young children without Clostridium difficile infection (CDI). These participants have no record of CDI diagnosis and serve as the control group to identify risk factors and biomarkers by comparing with the case group.

SUMMARY:
This study aims to investigate the epidemiological characteristics and biomarkers of Clostridium difficile infection in infants . By analyzing historical medical data and patient questionnaires, this retrospective cohort study will identify potential high-risk factors and establish baseline biomarkers to improve diagnosis and treatment for affected patients.

DETAILED DESCRIPTION:
This retrospective cohort study focuses on Clostridium difficile infection (CDI) in infants n, a relatively rare infection. The study will utilize data from hospital and community to identify the prevalence, risk factors, and unique biomarkers associated with CDI in pediatric patients. Key objectives include: (1) analyzing demographic and clinical characteristics of affected patients, (2) evaluating the high-risk factors of CDI, and (3) identifying biomarkers that can aid in early detection and treatment planning. Findings from this study are expected to contribute to the improvement of CDI management in pediatric care.

ELIGIBILITY:
Inclusion Criteria:

* Infants ( aged 0-2 years). Medical records and patient questionnaires available with confirmed Clostridium difficile infection (for case group) or without infection (for control group).

Exclusion Criteria:

* Infants beyond the age of 2 years at the time of diagnosis. Incomplete medical records or missing essential information related to infection status, feeding methods, or antibiotic exposure.Patients with other severe gastrointestinal conditions that may confound results.

Ages: 0 Months to 24 Months | Sex: All
Age Groups: Child
Study Population: Infants diagnosed with Clostridium difficile infection, along with age-matched control subjects without infection, recruited from affiliated hospitals and society. Participants will be selected based on inclusion and exclusion criteria to ensure a representative sample for studying infection risk factors and biomarker discovery in this population
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Infants With Identified High-Risk Factors for Clostridium difficile Infection (CDI) | Retrospective data review spanning from initial exposure to Clostridium difficile infection up to 12 months post-diagnosis.
  This measure reports the number of infants with high-risk factors associated with Clostridium difficile infection (CDI), as assessed by data on feeding methods, antibiotic use, and environmental exposures. Quantitative data will be analyzed to identify correlations and trends.

SECONDARY OUTCOMES:
Number of Identified Biomarkers Associated With Clostridium difficile Infection in Infants | From the initiation of the study until 12 months after the last sample collection
  This measure reports the number of specific biomarkers identified from collected biological samples that are associated with Clostridium difficile infection in infants and young children. Biomarkers include bacterial taxa, metabolites, and other biological indicators relevant to infection susceptibility and disease progression. These biomarkers will be analyzed to evaluate their potential roles as risk factors, diagnostic indicators, and predictors of disease outcomes.
Validation of Experimental Mouse Model for Clostridium difficile Infection and Biomarker Identification | From the initiation of the study until completion of biomarker identification, approximately 18 months
  This measure involves the validation of an experimental mouse model designed to simulate Clostridium difficile infection and identify key biomarkers associated with infection risk in infants. The validation process includes assessing the mouse model's effectiveness in replicating human disease conditions, such as microbiota composition and immune response. Specific biomarkers, including bacterial taxa, host immune markers, and metabolites, will be analyzed to evaluate the model's relevance for further biomarker discovery and translational research.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China, China

IPD SHARING:
Plan to Share IPD: No